CLINICAL TRIAL: NCT06526221
Title: Evaluating Urine Isoniazid Testing for Tuberculosis Disease in India to Detect Medication Nonadherence and Improve Treatment Outcomes
Brief Title: Evaluating Urine Isoniazid Testing to Detect Nonadherence to Tuberculosis Medications in India
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Tuberculosis Research Centre, India (Other Government); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00004944
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-07

CONDITIONS: Tuberculosis, Pulmonary; Medication Adherence
MeSH Terms: conditions — Tuberculosis, Pulmonary; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Based on NIH definitions, this is considered a clinical trial given that there is prospective assignment of an intervention (i.e., urine isoniazid testing) to evaluate medication adherence. As such, this could be considered a single group/arm study with prospective assignment of the intervention to all study participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Urine isoniazid testing (intervention arm) (Experimental): This is the only study group/arm in this study. Participants in this study arm will receive urine isoniazid testing using the IsoScreen test in the TB clinic at monthly clinical and medication refill visits at month 1, 2, 3, 4, and 5 (5 times total). The will also undergo urine isoniazid testing using the IsoScreen test at home visits after months 1, 3, and 5 of treatment (3 times total).
  Interventions: Diagnostic Test: Urine isoniazid testing (IsoScreen test)

INTERVENTIONS:
Diagnostic Test: Urine isoniazid testing (IsoScreen test) — Developed by Arkansas' Public Health Service in the 1970s, this test detects metabolites of isoniazid, a drug present in drug-susceptible TB regimens. IsoScreen (GFC Diagnostics, UK) is a commercial version of the Arkansas method with reagents enclosed in a plastic vial, into which 2mL of urine can be injected with a syringe. If the urine contains isoniazid, reagents turn purple/blue (suggesting a dose was taken in the last 24 hours or appropriate adherence) or green (suggesting a dose was taken 24-48 hours before or one missed dose). A yellow result (no color change) suggests medication has not been taken for >48 hours (two or more missed doses).

SUMMARY:
Tuberculosis (TB) is the leading infectious cause of death globally. India has the largest TB epidemic, accounting for one-quarter of cases and one-third of TB deaths worldwide. Nonadherence to medications is a central challenge in TB care leading to increased death, disease recurrence, and drug resistance. Despite its importance, detecting nonadherence in routine care is challenging, as current measurement approaches are inaccurate, not person-centered, or ineffective at improving outcomes. Early and accurate detection of nonadherence may serve as an entry point for differentiated care, in which people with TB at risk for poor outcomes can be given intensified interventions. Urine isoniazid testing is a validated, low-cost, point-of-care, and direct adherence measure that may be predictive of TB outcomes and therefore serve as an ideal triage test to enable differentiated care. However, to integrate urine testing into routine care, research is needed to: (1) understand how the test performs at scheduled clinic visits, (2) gain a rich understanding of root causes of nonadherence to better leverage urine test results, and (3) identify barriers and facilitators to implementation. In this study, the investigators propose conducting a 900 participant prospective cohort study with translational research involving clinical, behavioral, and implementation science to facilitate integration of urine isoniazid testing into India's national TB program. The investigators' central hypothesis is that urine testing can be integrated into routine care to facilitate early and accurate identification of people with TB who are likely to suffer poor outcomes, including death and TB recurrence. In Aim 1, the investigators will assess the accuracy of urine test results assessed at scheduled clinic visits in comparison to those assessed at unannounced home visits. In Aim 2, the investigators will assess the relationship between nonadherence detected by urine testing and subsequent unfavorable TB outcomes of death, loss to follow-up, treatment failure, and post-treatment TB recurrence.. This study proposal aims to develop an innovative but pragmatic strategy for early identification of TB medication nonadherence that is feasible in low- and middle-income countries with a high TB burden.

DETAILED DESCRIPTION:
Tuberculosis (TB) is the leading infectious cause of death globally. India has the largest TB epidemic, accounting for one-quarter of cases and one-third of global TB deaths. Nonadherence to TB medications is associated with increased death, TB recurrence, and drug resistance. Specifically, missing >10% of doses is associated with six times greater risk of poor TB outcomes.2 The association between nonadherence to TB medications and emergence of drug resistance is one of the most concerning from a public health perspective. For example, one study found that nonadherence to TB therapy was associated with independent elevated risk of acquiring drug resistance (adjusted odds ratio 19.7, 95%CI 1.7-234). Another study found that, among people being treated for multidrug-resistant (MDR) TB, each additional month in which a patient failed to take 80% of their prescribed medication doses was associated with elevated risk of developing extensively drug-resistant (XDR) TB (adjusted hazard ratio 1.2, 95% CI 1.01-1.4).

Despite its importance, detecting nonadherence in routine care is challenging, especially as TB programs in low- and middle-income countries (LMICs) have moved away from directly observed therapy. Our research shows indirect measures-e.g., cellphone-based technology, pill counts, and patient-reported measures-miss detecting >30% of people with TB who are nonadherent by urine isoniazid testing.

Urine isoniazid testing is a low-cost, validated, direct point-of-care adherence measure that is predictive of TB outcomes. In a 650-participant cohort study in India, one unannounced home visit was conducted for each participant during TB therapy to conduct urine testing. That study found: (1) nonadherence was common by urine testing, with 18% of participants having missed more than 1 dose, and (2) negative urine test results were associated with 3.9 increased odds of death and 3.8 increased odds of loss to follow-up from treatment.

While urine testing has benefits, further research is needed to evaluate its uses under TB programs setting First, urine testing may perform differently in clinic as compared to unannounced home visits, as people with TB may modify adherence behavior in anticipation of scheduled clinic visits. Research is needed to understand how well testing at clinic visits represents adherence and predicts TB outcomes. Second, research is needed to understand reasons for nonadherence (i.e., negative urine test results) to inform personalized interventions for differentiated care. Third, implementation science research is needed to evaluate the use of urine testing in routine care in a manner that could lead to sustained use and impact.

The investigators propose conducting translational research involving clinical, behavioural, and implementation science to evaluate the use of urine isoniazid testing in the TB program. The investigators' central hypothesis is that urine testing could be useful within the routine care to facilitate early and accurate identification of people with TB who are likely to suffer poor outcomes, including death and TB recurrence. If this hypothesis is correct, the urine assay could serve as a triage test for developing differentiated care strategies, in which people at risk for poor outcomes are identified early and given intensified care

The investigators have the following specific aims:

Aim 1. To assess the agreement between urine test results collected at prescheduled clinic in comparison to unannounced home visits.

Summary of this aim: The investigators will enroll a cohort of 900 people starting 6-month drug-susceptible TB therapy. For each participant, to enable comparison of clinic and home samples, the investigators will conduct 1 urine test at a scheduled clinic visit and 1 urine test at an unannounced home visit during each of the intensive (first 2 months), early continuation (second 2 months), and late continuation (last 2 months) treatment phases.

Aim 2. To assess the relationship between nonadherence by urine testing and subsequent TB outcomes.

Summary of this aim: The investigators will follow the Aim 1 cohort participants through the completion of TB treatment (which usually takes 6 months) and then for 12 months after treatment and assess the following unfavorable outcomes: death, treatment failure, loss to follow-up, and TB recurrence. The investigators will assess the association between nonadherence by urine testing (separately for clinic and home samples) and the composite of these unfavorable outcomes (primary outcome) and with each unfavorable outcome individually (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

1. 18+ years of age,
2. presumed or confirmed drug-susceptible pulmonary TB (with or without a previous TB history), and
3. taking an isoniazid-containing TB regimen.

Exclusion Criteria:

1. inability to provide informed consent, or
2. drug-resistant TB diagnosis or switch to another non-isoniazid-containing regimen (Note that this second exclusion criteria may result in retrospective exclusion from the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants experiencing a composite unfavorable tuberculosis treatment outcome | This outcome will be assessed during the course of TB treatment (usually about 6 months) and for the 12 months after TB treatment completion.
  The primary outcome will comprise the composite of: (1) loss to follow-up during treatment, (2) treatment failure, (3) death during the on-treatment or post-treatment period, and (4) TB recurrence. This will be reported as the number and proportion of participants experiencing one of the unfavorable outcomes, among all participants enrolled in the cohort study.

SECONDARY OUTCOMES:
The proportion of participants lost to follow-up during tuberculosis treatment | This outcome will be assessed during the course of TB treatment (usually about 6 months).
  This outcome will be defined as treatment interruption or being unable to contact a participant for >4 weeks. This will be reported as the number and proportion of participants experiencing loss to follow-up, among all participants enrolled in the cohort study.
The proportion of participants experiencing treatment failure (i.e., failure of tuberculosis treatment) | This outcome will be assessed during the course of TB treatment (usually about 6 months).
  A participant (person with TB) whose sputum smear or culture is positive at month 5 or later during treatment. This will be reported as the number and proportion of all participants experiencing treatment failure, among all participants enrolled in the cohort study.
The proportion of participants experiencing death | his outcome will be assessed during the course of TB treatment (usually about 6 months) and for the 12 months after TB treatment completion.
  Mortality from any cause. This will be reported as the number and proportion of participants experiencing death, among all participants enrolled in the cohort study.
The proportion of participants experiencing tuberculosis recurrence | This outcome will be assessed during the 12 months after completion of tuberculosis treamtent.
  Among study participants who achieved tuberculosis treatment completion, this will be defined as a positive sputum culture or an empirical (clinical) diagnosis of TB by healthcare providers in India's National TB Elimination Programme during the 12 months after a participant completed tuberculosis treatment. This will be reported as the number and proportion of participants experiencing TB recurrence, among all participants enrolled in the cohort study who completed TB treatment.

IPD SHARING:
Plan to Share IPD: Yes
Tuberculosis (TB) adherence and outcomes quantitative dataset: This will comprise one quantitative dataset of de-identified individual study participant data from 900 people with TB on treatment, including all quantitative data for the Aim 1 and Aim 2 cohort study. These data will be captured and stored as a Microsoft Excel CSV (comma-separated delimited text) file that can be uploaded into most statistical programs for analysis. As this dataset will be de-identified, individual-level data will be shared publicly through the NIAID Clinical Trials Data Repository (AccessClinicalData@NIAID).
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be made available as soon as possible or at the time of associated publication, whichever comes first.
Access Criteria: The NIAID Clinical Trials Data Repository provides metadata, persistent identifiers (i.e., digital object identifier), and long-term access. This repository is supported by the National Institute of Allergy and Infectious Diseases and datasets are available under a data access request process.